CLINICAL TRIAL: NCT03864003
Title: Community Health Workers and Teleaudiology as a Culturally-relevant Approach to Improving Access to Hearing Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Laura Coco, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1F32DC017081 (NIH)
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Community Health Workers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants randomized to the experimental group will receive hearing aid fitting and verification services via teleaudiology with local, hands-on support from a Community Health Worker.
  Interventions: Behavioral: Community Health Workers and Teleaudiology as a Culturally-Relevant Approach to Improving Access to Hearing Health Care
- Control Group (Active Comparator): Participants randomized to the control group will receive hearing aid fitting and verification services via teleaudiology with local, hands-on support from a non-Community Health Worker (undergraduate student in Speech, Language, and Hearing Sciences).
  Interventions: Behavioral: Community Health Workers and Teleaudiology as a Culturally-Relevant Approach to Improving Access to Hearing Health Care

INTERVENTIONS:
Behavioral: Community Health Workers and Teleaudiology as a Culturally-Relevant Approach to Improving Access to Hearing Health Care — In this project, remote hearing aid fittings will be delivered by an audiologist with patient-site support from a local facilitator for a cohort of older adults (>50 years) from a rural area that has been identified as under-resourced for hearing health care.

SUMMARY:
The purpose of this study is to test the feasibility of a teleaudiology intervention with assistance from Community Health Workers to improve access to hearing health care.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral hearing loss within the fitting range of study hearing aids

Exclusion Criteria:

* Medically unqualified to receive hearing aids
* Current hearing aid user
* Cognitively impaired

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Self-efficacy: The Self-Efficacy for Situational Communication Management Questionnaire | Baseline, 2 weeks, 6 weeks, and 12 weeks after hearing aid fitting
  The Self-Efficacy for Situational Communication Management Questionnaire (Jennings, 2005; Jennings et al, 2014) measures self-perceived hearing ability and hearing self-efficacy, or a participant's beliefs in their ability to manage communication with acquired hearing loss. The SESMQ contains 20 situations that are rated on two scales, hearing ability and perceived self-efficacy. Participants respond on a Likert scale from 0 (not well at all) to 10 (very well) to how well they can hear and how well they can manage in each situation. Total scores on each scale range from 0-200, with higher scores representing better perceived self-efficacy and better hearing ability. The two scales are scored and reported separately.
  We will evaluate the differences in SESMQ scores between experimental and control groups at 2-weeks post hearing aid fitting. Analyses will utilize baseline data and follow-up analyses will occur for 6-week and 12-week timepoints.

SECONDARY OUTCOMES:
Hearing aid benefit | Baseline, 6 weeks, and 14 weeks after hearing aid fitting
  The Effectiveness of Auditory Rehabilitation (Yueh et al., 2005; EAR) is a subjective scale of hearing aid function and quality of life. The first set of questions is administered before and after the hearing aid fitting, and relates to hearing concerns, including listening in quiet and other situations. The second set of questions relates to functioning with the hearing device, such as fit and convenience, and is administered after the hearing aid fitting.
  We will evaluate the differences in inner EAR scores between experimental and control groups at 6-weeks post hearing aid fitting. Analyses will utilize baseline data where appropriate and follow-up analyses will occur for 6-week and 12-week timepoints.
  Participants are asked to respond to statements on a five-point scale (i.e. very poor, poor, so-so, good, very good). Each answer is awarded a point. Higher cumulative scores indicate better benefit.
Satisfaction with teleaudiology service delivery | 2 weeks after hearing aid fitting
  Telehealth Satisfaction Scale (TeSS)
  The TeSS is a 10-item scale probing satisfaction with telehealth services. Responses are on a 4-point likert scale (Excellent, good, poor, fair). Higher cumulative scores represent better satisfaction.
Qualitative outcomes via semi-structured interviews | 14 weeks after hearing aid fitting
  Qualitative outcomes will target participants' subjective experience on access to hearing health care, self-efficacy, benefit, and satisfaction with service delivery and hearing aids.
Average hours of hearing aid usage per day | 2 weeks, 6 weeks, 14 weeks after hearing aid fitting
  We will ask participants the approximate average hours per day they use their hearing aid. This information will also be collected from the hearing aid programming software.
Subjective hearing aid benefit | 2 weeks, 6 weeks, 14 weeks after hearing aid fitting
  Subjective hearing aid benefit will also be measured using a patient reported outcome measure, the International Outcome Inventory for Hearing Aids (IOI-HA). Participants are asked to respond to seven questions on their experience with their hearing aids. Questions on the IOI-HA are on a 5-point Likert-type scale. Cumulative scores range from zero to 35. Higher scores represent better benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Coco, AuD, Principal Investigator — University of Arizona
Locations (1):
- Mariposa Community Health Center, Nogales, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coco L, Leon K, Navarro C, Piper R, Carvajal S, Marrone N. "Close to My Community": A Qualitative Study of Community Health Worker-Supported Teleaudiology Hearing Aid Services. Ear Hear. 2024 Sep-Oct 01;45(5):1191-1201. doi: 10.1097/AUD.0000000000001507. Epub 2024 May 30. PMID 38812073
- [Derived] Marrone NL, Nieman CL, Coco L. Community-Based Participatory Research and Human-Centered Design Principles to Advance Hearing Health Equity. Ear Hear. 2022 Jul-Aug 01;43(Suppl 1):33S-44S. doi: 10.1097/AUD.0000000000001183. Epub 2020 Jun 13. PMID 35724253